CLINICAL TRIAL: NCT06850740
Title: The Efficacy of Co-Spinal Ondansetron In Inguinal Herniorrhaphy: A Randomized Controlled Trial
Brief Title: Efficacy of Co-Spinal Ondansetron In Inguinal Herniorrhaphy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, assistant professor, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Co ondansetrone
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Ondansetron; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetrone (Active Comparator): will receive 8 mg of ondansetron (ZOFATRONE®, 8 mg/4 mL, EVA Pharma, Egypt) over 100 ml of normal saline solution over 10 minutes, starting with skin preparation for spinal anesthesia via the intravenous axis and a rapid intravenous (IV) infusion of 15 mL/kg of Ringer's solution that will be co-loaded during spinal anesthesia.
  Interventions: Drug: Ondansetron 8mg
- Saline (Placebo Comparator): will be managed by administering 100 ml of normal saline solution over 10 minutes, starting with the skin preparation for spinal anesthesia via the intravenous axis and a rapid intravenous (IV) infusion of 15 mL/kg of Ringer's solution that will be co-loaded during spinal anesthesia.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ondansetron 8mg — Patients will receive 8 mg of ondansetron (ZOFATRONE®, 8 mg/4 mL, EVA Pharma, Egypt)
  Other Names: OND
  Arms: Ondansetrone
Drug: Normal Saline — Patients will be managed by administering 100 ml of normal saline solution as placebo
  Other Names: Saline
  Arms: Saline

SUMMARY:
Ondansetron, a selective serotonin 5-HT3 receptor antagonist, is well known for its antiemetic effects. However, its ability to reduce hypotension during spinal anesthesia has recently sparked great interest. In clinical practice, administering ondansetron before spinal anesthesia has produced promising results.

DETAILED DESCRIPTION:
This prospective randomized double-blinded controlled study will be conducted on 46 patients undergoing inguinal herniorrhaphy at Suez Canal University Hospital and will be randomly assigned to one of the two groups using a table of random numbers. Group A (23 patients) will be administered 8 mg of ondansetron diluted in 100 ml of normal saline, starting with the skin preparation for spinal anesthesia through the intravenous axis to be finished in 10 minutes. Group B (23 patients) will be administered 100 ml of normal saline, starting with the skin preparation for spinal anesthesia through the intravenous axis, to be finished in 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for inguinal herniorrhaphy in Suez Canal University Hospitals
* Height: 150 to 180 cm.
* Body mass index (BMI): not more than 35 kg/m².
* Patients are ASA I (American Society of Anesthesiology physical status Grade I) = (normal healthy patients), ASA II (American Society of Anesthesiologists physical status Grade II) = (patients with mild systemic disease and no functional limitations).

Exclusion Criteria:

* Patients refused to participate in the study.
* Contraindications of spinal anesthesia.
* Known allergy to bupivacaine or ondansetron.
* Patients with a history of arrhythmia, especially those with prolonged QT intervals.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Ephedrine | From the time of spinal anaesthesia administration till the end of surgery not exceeding two hors
  Total intraoperative ephedrine consumption.

SECONDARY OUTCOMES:
Nausea and vomiting | From the time of end of surgery till the pass of the first 24 hours postoperatively
  Incidence of post operative nausea and vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt